CLINICAL TRIAL: NCT00513396
Title: A Randomized Control Trial Of High-Dose Isoniazid Adjuvant Therapy For Multidrug Resistant Tuberculosis
Brief Title: High-Dose Isoniazid Adjuvant Therapy for Multidrug Resistant Tuberculosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: GSVM Medical College (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TB chest - 1/2005
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Last update posted 2007-08-08 (Estimated); Status verified 2007-07

CONDITIONS: Tuberculosis, Multidrug-Resistant
Keywords: Randomized control trial; multidrug resistant tuberculosis; isoniazid; standardized regimen; adjuvant therapy
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant | interventions — Isoniazid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Isoniazid
- 2 (Active Comparator)
  Interventions: Drug: Isoniazid
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Isoniazid — High-dose isoniazid (16-18 mg/kg/day) in addition to standardized regimen that included the following: kanamycin (15 mg/kg/day), levofloxacin (7.5-15 mg/kg/day), protionamide (10-20 mg/kg/day), cycloserine (10-20 mg/kg/day) and p-aminosalicylic acid (150 mg/kg/day)
  Regular dose isoniazid (5 mg/kg/day) in addition to standard regimen that included the following: kanamycin (15 mg/kg/day), levofloxacin (7.5-15 mg/kg/day), protionamide (10-20 mg/kg/day), cycloserine (10-20 mg/kg/day) and p-aminosalicylic acid (150 mg/kg/day)
  Arms: 1; 2
Drug: Placebo — Similar appearing and similarly packaged placebo tablets in addition to the standardized regimen that included the following: kanamycin (15 mg/kg/day), levofloxacin (7.5-15 mg/kg/day), protionamide (10-20 mg/kg/day), cycloserine (10-20 mg/kg/day) and p-aminosalicylic acid (150 mg/kg/day)
  Arms: 3

SUMMARY:
The need for a standardized treatment protocol for multidrug resistant tuberculosis (MDR-TB) in resource-limited countries is being increasingly recognized. This single center, double blind, randomized controlled trial was designed to compare the time required for sputum culture conversion and extent of radiological improvement in cases of MDR pulmonary tuberculosis when isoniazid was included (both at a regular dose and at a high dose) as an adjuvant to the standardized second line of treatment. The study was designed to test the hypothesis that inclusion of high-dose isoniazid will enhance the effectiveness of the second line of treatment in cases of MDR-TB without significantly increasing the toxicity.

DETAILED DESCRIPTION:
Tuberculosis was declared a global emergency by the World Health Organization (WHO) in 1993. The global problem of tuberculosis is further complicated by a substantial increase in drug resistant tuberculosis. Available data suggest that drug resistant TB especially multi drug resistant may represent a public health threat in areas with a high prevalence of tuberculosis, suboptimal TB control programmes and/ or HIV. The cure rate of these cases has been reported to be lower than for non-drug resistant TB with a failure rate of 44%. New therapies for MDR-TB have not been introduced since the fluoroquinolones in the 1970s. Strains of Mycobacterium Tuberculosis (M. tub.) in H resistant cases often contain mixture of susceptible & resistant organisms. Use of high dose H (16- 20 mg/kg) can eliminate susceptible & those with low level resistance4. This Study was done to evaluate the role of isoniazid (INH) at high & normal dosages as an adjuvant therapy in treatment of patients with persistent culture positive pulmonary tuberculosis despite 6 months of continuous first line antitubercular treatment and on culture at least resistant to isoniazid and rifampicin.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients reporting to the study center
* Sputum-positive for acid-fast bacilli
* HIV-uninfected
* MDR-TB defined as resistance to at least the following two drugs: Isoniazid and Rifampicin.

Exclusion Criteria:

* Unwilling to give consent
* Abnormal renal or hepatic profile
* History suggestive of isoniazid hypersensitivity
* Pregnancy
* Lactating mother
* Previous history of taking any of the following: kanamycin, prothionamide, levofloxacin, cycloserine and p-aminosalicylic acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2004-01; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Time to sputum culture conversion | 1 year

SECONDARY OUTCOMES:
Extent of radiological improvement | 1 year
Proportion with peripheral neuropathy | 1 year
Proportion with hepatotoxicity | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Subodh Katiyar, MD, Study Chair — GSVM Medical College, Kanpur, India; Shivesh Prakash, MBBS, Principal Investigator — GSVM Medical College, Kanpur, India; Shailesh Bihari, MD, Principal Investigator — GSVM Medical College, Kanpur, India; Hemant Kulkarni, MD, Principal Investigator — Lata Medical Research Foundation, Nagpur, India; Manju Mamtani, MD, Principal Investigator — Lata Medical Research Foundation, Nagpur, India